CLINICAL TRIAL: NCT04502251
Title: Association of Low Doses of Naltrexone and Transcranial Direct Current Stimulation in Fibromyalgia: Randomized Clinical Trial, Blind, Controlled With Placebo
Brief Title: LDN and tDCS in Fibromyalgia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centro Universitario La Salle (Other)
Collaborators: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Andressa de Souza, Principal Investigator, Centro Universitario La Salle
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 70005317.5.0000.5307
Record Dates: First submitted 2020-07-25; First posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Fibromyalgia
Keywords: tDCS; LDN; Transcranial Direct Current Stimulation; Low Dose Naltrexone
MeSH Terms: conditions — Fibromyalgia | interventions — Naltrexone; Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: A randomized, double-blinded, parallel, controlled with placebo and sham stimulation, clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blinded study, in which the participants and the outcomes assessor, who is the same as the investigator and the care provider, are blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- LDN + tDCS (Active Comparator): Low Dose Naltrexone and Transcranial Direct Current Stimulation
  Interventions: Drug: Low-Dose Naltrexone; Device: Transcranial Direct Current Stimulation
- LDN + Sham tDCS (Sham Comparator): Low Dose Naltrexone and Sham Transcranial Direct Current Stimulation
  Interventions: Drug: Low-Dose Naltrexone; Device: Sham Transcranial Direct Current Stimulation
- Placebo + tDCS (Placebo Comparator): Placebo and Transcranial Direct Current Stimulation
  Interventions: Device: Transcranial Direct Current Stimulation; Drug: Placebo
- Placebo + Sham tDCS (Other): Placebo and Sham Transcranial Direct Current Stimulation
  Interventions: Drug: Placebo; Device: Sham Transcranial Direct Current Stimulation

INTERVENTIONS:
Drug: Low-Dose Naltrexone — 4.5mg daily dose, orally, during 26 days
  Other Names: LDN
  Arms: LDN + Sham tDCS; LDN + tDCS
Device: Transcranial Direct Current Stimulation — An anodal electrode was placed on the scalp above the primary motor cortex (M1), contralateral to the dominant cortex. The cathodal electrode was placed on the supraorbital contralateral area. The current used was 2mA during 20 minutes.
  Other Names: tDCS
  Arms: LDN + tDCS; Placebo + tDCS
Drug: Placebo — The capsule presented the same format, size and color as LDN capsules, however the excipient used was starch.
  Arms: Placebo + Sham tDCS; Placebo + tDCS
Device: Sham Transcranial Direct Current Stimulation — Sham-tDCS stimulation consists of an active current during 30 seconds
  Other Names: Sham tDCS
  Arms: LDN + Sham tDCS; Placebo + Sham tDCS

SUMMARY:
Fibromyalgia is a complex generalized and diffuse musculoskeletal chronic pain; and pharmacological approaches are widely used to relieve pain and increase life quality. In this context, low-dose naltrexone (LDN) was able to increase nociceptive threshold in patients with fibromyalgia. Moreover, non-pharmacological techniques, like Transcranial Direct Current Stimulation (tDCS), have been shown effective for pain management. This study aims to evaluate the analgesic and neuromodulatory effect of combined LDN followed by tDCS in fibromyalgia patients. This is a randomized, double-blinded, parallel, placebo/sham-controlled trial, in which 92 (10% loss) women with fibromyalgia will be included included and signed the informed consent. Patients will be allocated into 4 groups: tDCS+LDN (n=21), Sham-tDCS+LDN (n=22), tDCS+Placebo (n=22), and Sham-tDCS+Placebo (n=21). LDN or placebo (p.o.) intervention lasts 26 days, in the last five, tDCS will be applied (sham or active, 20min, 2mA). Questionnaires assessed are: Sociodemographic, Visual Analog Pain Scale (VAS), Pain Catastrophizing Scale (PCS), State-Trait Anxiety Inventory (STAI), Fibromyalgia Impact Questionnaire (FIQ), Beck Depression Inventory (BDI-II), Chronic Pain Profile Scale (CPP). Also, pain measures were taken: Pain Pressure Threshold (PPT) and Conditioned Pain Modulation (CPM). Blood samples will be collected to analyze Brain Derived Neurotrophic Factor (BDNF) serum levels.

ELIGIBILITY:
Inclusion Criteria:

* signed the consent form
* women from 18 to 65 years
* confirmed diagnosis of fibromyalgia according 2016 American College of Rheumatology criteria
* read and write
* pain higher than 6 in the Visual Analogue Scale (VAS), in the last 3 months
* chronic stable treatment in the last 3 months.

Exclusion Criteria:

* in use of opioid drugs;
* pregnancy or not using anticontraceptive
* history of alcohol or drug abuse in the last 6 months
* history of neurological pathologies
* history of arrhythmia
* history of use of drugs that might change vascular response
* history of head trauma
* history of neurosurgery
* decompensated systemic diseases or chronic inflammatory diseases (lupus, rheumatoid arthritis, Sjogren syndrome, Reiter syndrome)
* history of non-compensated hypothyroidism
* personal history of cancer.

Ages: 8 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Pain in VAS | Change between baseline and after association (26 days from baseline)
  Visual Analogue Scale (VAS) that goes from 0 cm (without pain) to 10cm (worst pain).

SECONDARY OUTCOMES:
Depressive symptoms | Change between baseline and after association (26 days from baseline)
  Beck Depression Inventory (BDI-II) that goes from 0 (without depressive symptoms) to 63 (worst depressive symptoms)
Anxiety levels | Change between baseline and after association (26 days from baseline)
  State-Trait Anxiety Inventory (STAI) divided into state anxiety (from 0 to 52, the higher the worse) and trait anxiety (from 0 to 48, the higher the worse)
Pain Catastrophizing Thought | Change between baseline and after association (26 days from baseline)
  Pain Catastrophizing Scale (PCS): divided into rumination (from 0 to 16, the higher the worse), magnification (from 0 to 12, the higher the worse) and hopelessness (from 0 to 24, the higher the worse). Total goes from 0 to 52, the higher the worse
Profile of Chronic Pain | Change between baseline and after association (26 days from baseline)
  Profile of Chronic Pain Scale (PCP:S): divided into Frequency and Intensity of Pain (from 0 to 30, the higher the worse), Pain Effect in Activities (from 0 to 36, the higher the worse) and Pain Effect in Emotions (from 0 to 25, the higher the worse)
Pain Pressure Threshold | Change between baseline and after association (26 days from baseline)
  Pain Pressure Threshold (PPT) measured using an electronic algometer applied in the right forearm; and patients need to report the first pain sensation (minimum pain) and maximum pain. Threshold goes from 0 to the maximum value the patient can hold, the higher the value, better is the result
Conditioned Pain Modulation | Change between baseline and after association (26 days from baseline)
  Conditioned Pain Modulation (CPM) with an algometer (PPT task), the patient informed when felt a pain equal to 6 in the VAS. This pain level was applied in the right forearm for 30 seconds, while the left forearm (non-dominant hand) was submerged in water from 0˚C to 1.5˚C; after 30s, patients reported their pain in each of the arms. CPM = left forearm VAS - 6. (from -4 to 6, the value must be as closest to -4 as possible, meaning the higher the worse)
Serum BDNF | Change between baseline and after association (26 days from baseline)
  Blood sample collected and centrifuged, the supernatant aliquoted for BDNF analysis using ELISA technique, according to manufacturer's instructions (values start in 0, patients with fibromyalgia usually have higher levels of serum BDNF, therefore the higher the worse)

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade La Salle, Canoas, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Clauw DJ. Fibromyalgia: a clinical review. JAMA. 2014 Apr 16;311(15):1547-55. doi: 10.1001/jama.2014.3266. PMID 24737367
- [Background] van Hecke O, Torrance N, Smith BH. Chronic pain epidemiology and its clinical relevance. Br J Anaesth. 2013 Jul;111(1):13-8. doi: 10.1093/bja/aet123. PMID 23794640
- [Background] Chapman CR, Nakamura Y. A passion of the soul: an introduction to pain for consciousness researchers. Conscious Cogn. 1999 Dec;8(4):391-422. doi: 10.1006/ccog.1999.0411. PMID 10600241
- [Background] Yunus MB. Fibromyalgia and overlapping disorders: the unifying concept of central sensitivity syndromes. Semin Arthritis Rheum. 2007 Jun;36(6):339-56. doi: 10.1016/j.semarthrit.2006.12.009. Epub 2007 Mar 13. PMID 17350675
- [Background] Burgmer M, Pogatzki-Zahn E, Gaubitz M, Wessoleck E, Heuft G, Pfleiderer B. Altered brain activity during pain processing in fibromyalgia. Neuroimage. 2009 Jan 15;44(2):502-8. doi: 10.1016/j.neuroimage.2008.09.008. Epub 2008 Sep 24. PMID 18848998
- [Background] Harris RE, Gracely RH, McLean SA, Williams DA, Giesecke T, Petzke F, Sen A, Clauw DJ. Comparison of clinical and evoked pain measures in fibromyalgia. J Pain. 2006 Jul;7(7):521-7. doi: 10.1016/j.jpain.2006.01.455. PMID 16814691
- [Background] Sluka KA, Clauw DJ. Neurobiology of fibromyalgia and chronic widespread pain. Neuroscience. 2016 Dec 3;338:114-129. doi: 10.1016/j.neuroscience.2016.06.006. Epub 2016 Jun 9. PMID 27291641
- [Background] Yunus MB. Central sensitivity syndromes: a new paradigm and group nosology for fibromyalgia and overlapping conditions, and the related issue of disease versus illness. Semin Arthritis Rheum. 2008 Jun;37(6):339-52. doi: 10.1016/j.semarthrit.2007.09.003. Epub 2008 Jan 14. PMID 18191990
- [Background] Lobo CP, Pfalzgraf AR, Giannetti V, Kanyongo G. Impact of invalidation and trust in physicians on health outcomes in fibromyalgia patients. Prim Care Companion CNS Disord. 2014 Oct 9;16(5):10.4088/PCC.14m01664. doi: 10.4088/PCC.14m01664. eCollection 2014. PMID 25667809
- [Background] Fitzcharles MA, Ste-Marie PA, Mailis A, Shir Y. Adjudication of fibromyalgia syndrome: challenges in the medicolegal arena. Pain Res Manag. 2014 Nov-Dec;19(6):287-92. doi: 10.1155/2014/742830. PMID 25479148
- [Background] Wolfe F, Smythe HA, Yunus MB, Bennett RM, Bombardier C, Goldenberg DL, Tugwell P, Campbell SM, Abeles M, Clark P, et al. The American College of Rheumatology 1990 Criteria for the Classification of Fibromyalgia. Report of the Multicenter Criteria Committee. Arthritis Rheum. 1990 Feb;33(2):160-72. doi: 10.1002/art.1780330203. PMID 2306288
- [Background] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Katz RS, Mease P, Russell AS, Russell IJ, Winfield JB, Yunus MB. The American College of Rheumatology preliminary diagnostic criteria for fibromyalgia and measurement of symptom severity. Arthritis Care Res (Hoboken). 2010 May;62(5):600-10. doi: 10.1002/acr.20140. PMID 20461783
- [Background] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Hauser W, Katz RL, Mease PJ, Russell AS, Russell IJ, Walitt B. 2016 Revisions to the 2010/2011 fibromyalgia diagnostic criteria. Semin Arthritis Rheum. 2016 Dec;46(3):319-329. doi: 10.1016/j.semarthrit.2016.08.012. Epub 2016 Aug 30. PMID 27916278
- [Background] Younger J, Noor N, McCue R, Mackey S. Low-dose naltrexone for the treatment of fibromyalgia: findings of a small, randomized, double-blind, placebo-controlled, counterbalanced, crossover trial assessing daily pain levels. Arthritis Rheum. 2013 Feb;65(2):529-38. doi: 10.1002/art.37734. PMID 23359310
- [Background] Parker CE, Nguyen TM, Segal D, MacDonald JK, Chande N. Low dose naltrexone for induction of remission in Crohn's disease. Cochrane Database Syst Rev. 2018 Apr 1;4(4):CD010410. doi: 10.1002/14651858.CD010410.pub3. PMID 29607497
- [Background] Brown N, Panksepp J. Low-dose naltrexone for disease prevention and quality of life. Med Hypotheses. 2009 Mar;72(3):333-7. doi: 10.1016/j.mehy.2008.06.048. Epub 2008 Nov 28. PMID 19041189
- [Background] Younger J, Parkitny L, McLain D. The use of low-dose naltrexone (LDN) as a novel anti-inflammatory treatment for chronic pain. Clin Rheumatol. 2014 Apr;33(4):451-9. doi: 10.1007/s10067-014-2517-2. Epub 2014 Feb 15. PMID 24526250
- [Background] Tempel A, Gardner EL, Zukin RS. Neurochemical and functional correlates of naltrexone-induced opiate receptor up-regulation. J Pharmacol Exp Ther. 1985 Feb;232(2):439-44. PMID 2982011
- [Background] Fregni F, Boggio PS, Lima MC, Ferreira MJ, Wagner T, Rigonatti SP, Castro AW, Souza DR, Riberto M, Freedman SD, Nitsche MA, Pascual-Leone A. A sham-controlled, phase II trial of transcranial direct current stimulation for the treatment of central pain in traumatic spinal cord injury. Pain. 2006 May;122(1-2):197-209. doi: 10.1016/j.pain.2006.02.023. Epub 2006 Mar 27. PMID 16564618
- [Background] Nitsche MA, Fricke K, Henschke U, Schlitterlau A, Liebetanz D, Lang N, Henning S, Tergau F, Paulus W. Pharmacological modulation of cortical excitability shifts induced by transcranial direct current stimulation in humans. J Physiol. 2003 Nov 15;553(Pt 1):293-301. doi: 10.1113/jphysiol.2003.049916. Epub 2003 Aug 29. PMID 12949224
- [Background] Nitsche MA, Schauenburg A, Lang N, Liebetanz D, Exner C, Paulus W, Tergau F. Facilitation of implicit motor learning by weak transcranial direct current stimulation of the primary motor cortex in the human. J Cogn Neurosci. 2003 May 15;15(4):619-26. doi: 10.1162/089892903321662994. PMID 12803972
- [Background] Fregni F, Boggio PS, Nitsche M, Bermpohl F, Antal A, Feredoes E, Marcolin MA, Rigonatti SP, Silva MT, Paulus W, Pascual-Leone A. Anodal transcranial direct current stimulation of prefrontal cortex enhances working memory. Exp Brain Res. 2005 Sep;166(1):23-30. doi: 10.1007/s00221-005-2334-6. Epub 2005 Jul 6. PMID 15999258
- [Background] Marlow NM, Bonilha HS, Short EB. Efficacy of transcranial direct current stimulation and repetitive transcranial magnetic stimulation for treating fibromyalgia syndrome: a systematic review. Pain Pract. 2013 Feb;13(2):131-45. doi: 10.1111/j.1533-2500.2012.00562.x. Epub 2012 May 28. PMID 22631436
- [Background] Zhu CE, Yu B, Zhang W, Chen WH, Qi Q, Miao Y. Effiectiveness and safety of transcranial direct current stimulation in fibromyalgia: A systematic review and meta-analysis. J Rehabil Med. 2017 Jan 19;49(1):2-9. doi: 10.2340/16501977-2179. PMID 27983739
- [Background] Boros K, Poreisz C, Munchau A, Paulus W, Nitsche MA. Premotor transcranial direct current stimulation (tDCS) affects primary motor excitability in humans. Eur J Neurosci. 2008 Mar;27(5):1292-300. doi: 10.1111/j.1460-9568.2008.06090.x. Epub 2008 Feb 29. PMID 18312584
- [Background] Fregni F, Gimenes R, Valle AC, Ferreira MJ, Rocha RR, Natalle L, Bravo R, Rigonatti SP, Freedman SD, Nitsche MA, Pascual-Leone A, Boggio PS. A randomized, sham-controlled, proof of principle study of transcranial direct current stimulation for the treatment of pain in fibromyalgia. Arthritis Rheum. 2006 Dec;54(12):3988-98. doi: 10.1002/art.22195. PMID 17133529
- [Background] Fagerlund AJ, Hansen OA, Aslaksen PM. Transcranial direct current stimulation as a treatment for patients with fibromyalgia: a randomized controlled trial. Pain. 2015 Jan;156(1):62-71. doi: 10.1016/j.pain.0000000000000006. PMID 25599302
- [Background] Wang YP, Gorenstein C. Psychometric properties of the Beck Depression Inventory-II: a comprehensive review. Braz J Psychiatry. 2013 Oct-Dec;35(4):416-31. doi: 10.1590/1516-4446-2012-1048. Epub 2013 Dec 23. PMID 24402217
- [Background] Kaipper MB, Chachamovich E, Hidalgo MP, Torres IL, Caumo W. Evaluation of the structure of Brazilian State-Trait Anxiety Inventory using a Rasch psychometric approach. J Psychosom Res. 2010 Mar;68(3):223-33. doi: 10.1016/j.jpsychores.2009.09.013. Epub 2009 Dec 9. PMID 20159207
- [Background] Caumo W, Ruehlman LS, Karoly P, Sehn F, Vidor LP, Dall-Agnol L, Chassot M, Torres IL. Cross-cultural adaptation and validation of the profile of chronic pain: screen for a Brazilian population. Pain Med. 2013 Jan;14(1):52-61. doi: 10.1111/j.1526-4637.2012.01528.x. Epub 2012 Nov 21. PMID 23171145
- [Background] Seoane-Mato D, Sanchez-Piedra C, Silva-Fernandez L, Sivera F, Blanco FJ, Perez Ruiz F, Juan-Mas A, Pego-Reigosa JM, Narvaez J, Quilis Marti N, Cortes Verdu R, Anton-Pages F, Quevedo Vila V, Garrido Courel L, Del Amo NDV, Paniagua Zudaire I, Anez Sturchio G, Medina Varo F, Ruiz Tudela MDM, Romero Perez A, Ballina J, Brandy Garcia A, Fabregas Canales D, Font Gaya T, Bordoy Ferrer C, Gonzalez Alvarez B, Casas Hernandez L, Alvarez Reyes F, Delgado Sanchez M, Martinez Dubois C, Sanchez-Fernandez SA, Rojas Vargas LM, Garcia Morales PV, Olive A, Rubio Munoz P, Larrosa M, Navarro Ricos N, Graell Martin E, Chamizo E, Chaves Chaparro L, Rojas Herrera S, Pons Dolset J, Polo Ostariz MA, Ruiz-Alejos Garrido S, Macia Villa C, Cruz Valenciano A, Gonzalez Gomez ML, Morcillo Valle M, Palma Sanchez D, Moreno Martinez MJ, Mayor Gonzalez M, Atxotegi Saenz de Buruaga J, Urionaguena Onaindia I, Blanco Caceres BA, Diaz-Gonzalez F, Bustabad S. Prevalence of rheumatic diseases in adult population in Spain (EPISER 2016 study): Aims and methodology. Reumatol Clin (Engl Ed). 2019 Mar-Apr;15(2):90-96. doi: 10.1016/j.reuma.2017.06.009. Epub 2017 Jul 31. English, Spanish. PMID 28774657
- [Background] Bernardy K, Klose P, Busch AJ, Choy EH, Hauser W. Cognitive behavioural therapies for fibromyalgia. Cochrane Database Syst Rev. 2013 Sep 10;2013(9):CD009796. doi: 10.1002/14651858.CD009796.pub2. PMID 24018611
- [Background] Younger J, Mackey S. Fibromyalgia symptoms are reduced by low-dose naltrexone: a pilot study. Pain Med. 2009 May-Jun;10(4):663-72. doi: 10.1111/j.1526-4637.2009.00613.x. Epub 2009 Apr 22. PMID 19453963
- [Background] Khedr EM, Omran EAH, Ismail NM, El-Hammady DH, Goma SH, Kotb H, Galal H, Osman AM, Farghaly HSM, Karim AA, Ahmed GA. Effects of transcranial direct current stimulation on pain, mood and serum endorphin level in the treatment of fibromyalgia: A double blinded, randomized clinical trial. Brain Stimul. 2017 Sep-Oct;10(5):893-901. doi: 10.1016/j.brs.2017.06.006. Epub 2017 Jun 23. PMID 28684258
- [Background] Boggio PS, Rigonatti SP, Ribeiro RB, Myczkowski ML, Nitsche MA, Pascual-Leone A, Fregni F. A randomized, double-blind clinical trial on the efficacy of cortical direct current stimulation for the treatment of major depression. Int J Neuropsychopharmacol. 2008 Mar;11(2):249-54. doi: 10.1017/S1461145707007833. Epub 2007 Jun 11. PMID 17559710

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-11-13): https://cdn.clinicaltrials.gov/large-docs/51/NCT04502251/Prot_SAP_ICF_000.pdf